CLINICAL TRIAL: NCT01092546
Title: A Principal, Prospective, Open-label Biopsy Study to Validate Detection of Cerebral Cortical Amyloid With Flutemetamol (18F) Injection in Normal Pressure Hydrocephalus (NPH) Subjects.
Brief Title: Positron Emission Tomography Imaging of Brain Amyloid in Normal Pressure Hydrocephalus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Changed focus of the program
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-067-009
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Amyloid; Normal pressure hydrocephalus (NPH); Positron Emission Tomography (PET); Standard uptake value ratios (SUVR)
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Alzheimer Disease | interventions — flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: [18F]Flutemetamol

INTERVENTIONS:
Drug: [18F]Flutemetamol — All subjects will receive an IV dose of [18F]flutemetamol (less than 10 mg flutemetamol). The nominal activity of a single administration of [18F]flutemetamol will be 185 MBq.
  Other Names: Flutemetamol; AH110690

SUMMARY:
To determine the level of association between the quantitative estimates of brain uptake of [18F]flutemetamol and the quantitative immunohistochemical and histochemistry estimates of amyloid levels in frontal lobe biopsy samples obtained from subjects during shunt placement for NPH.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 50 years of age.
* The subjects' general health is adequate to comply with study procedures.
* The subject has been scheduled for a shunt placement procedure for the treatment of NPH.

Exclusion Criteria:

* The subject has a contraindication for MRI or PET.
* The subject is pregnant or lactating.
* The subject has a known or suspected hypersensitivity/allergy to [18F]flutemetamol or to any of the excipients.
* The subject has participated in any clinical study using an investigational agent within 30 days of dosing.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Mansfield, MS, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Started with 16 subjects and 4 withdrew prior to dosing leaving 12 subjects for study.
Groups:
- Arm 1-Flutemetamol Injection: [18F]Flutemetamol : All subjects received an IV dose of [18F]flutemetamol (less than 10 mg flutemetamol). The nominal activity of a single administration of [18F]flutemetamol will be 185 MBq.
Period: Overall Study
Arm/Group | Arm 1-Flutemetamol Injection
Started | 16
Completed | 12
Not Completed | 4
Not completed — Subjects withdrawn prior to dosing | 4

BASELINE CHARACTERISTICS:
Population: 4 of the 16 Subjects were withdrawn prior to study dosing.
Groups:
- Arm 1-Flutemetamol Injection: [18F]Flutemetamol : All subjects will receive an IV dose of [18F]flutemetamol (less than 10 mg flutemetamol). The nominal activity of a single administration of [18F]flutemetamol will be 185 MBq.
Arm/Group | Arm 1-Flutemetamol Injection
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Standard Uptake Value Ratio (SUVR) at the Site of the Biopsy Based on the "Cerebellum" (CER) as the Reference Region.
Description: The level of association between the quantitative estimates of brain uptake of [18F]flutemetamol and the quantitative immunohistochemical estimates of amyloid levels in biopsy samples obtained during shunt placement in patients who have Normal Pressure Hydrocephalus (NPH). The quantitative estimates of brain uptake of [18F]flutemetamol (SUVR) will be made from the analysis of PET images.
Time Frame: Post flutemetamol Injection
Population: The correlation coefficient listed in the table is between SUVR-CER and the percent area of Amyloid.
  Stain IHC 4G8 was used as the Standard of Truth. Standard Uptake Value Ratio (SUVR) at the site of the biopsy was based on the cerebullum (CER) as the reference region.
Measure: Number; unit: Correlation Coefficient of the Site
Arm/Group | Arm 1-Flutemetamol Injection
Number analyzed (Participants) | 12
Correlation Coefficient of the Site
  Biopsy Site | 0.64
  Contralateral to Biopsy Site | 0.69
  Composite Region | 0.81

2. Secondary Outcome: Standard Uptake Value Ratio (SUVR) at the Site of the Biopsy Based on the "Pons" as the Reference Region.
Description: The level of association between SUVR and the quantitative estimates (area percents) of amyloid levels for the following regions: Biopsy site and Contralateral and Composite Regions.
Time Frame: Post flutemetamol administration
Population: The correlation coefficient listed in the table is between SUVR-Pons and the percent area of Amyloid.
  Stain IHC 4G8 was used as the Standard of Truth. Standard Uptake Value Ratio (SUVR) at the site of the biopsy was based on the Pons as the reference region.
Measure: Number; unit: Correlation Coefficient of the site
Arm/Group | Arm 1-Flutemetamol Injection
Number analyzed (Participants) | 12
Correlation Coefficient of the site
  Biopsy Site | 0.60
  Contralateral to Biopsy Site | 0.63
  Composite Region | 0.76

ADVERSE EVENTS:
Arm/Group | Arm 1-Flutemetamol Injection
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No